CLINICAL TRIAL: NCT05118659
Title: Mulligan Therapy Effects In Healthy Subjects With Induced Vertigo. A Randomized And Controlled Clinic Study
Brief Title: Mulligan Therapy Effects In Healthy Subjects With Induced Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitario La Salle (Other)
Responsible Party: Principal Investigator, Jose Vicente Leon Hernandez, Principal Investigator, Centro Universitario La Salle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CSEULS-PI-198/2018
Record Dates: First submitted 2021-10-19; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SNAG GROUP (Experimental): The SNAG group received a treatment based on sustained apophyseal glides in a postero-anterior direction on C2 with a dose of three series of ten repetitions each, combined with active cervical extension.
  Interventions: Procedure: sustained natural apophyseal glides
- SHAM SNAG GROUP (Sham Comparator): The placebo SNAG group received a simulation of the contact used for the SNAGs, without any vertebral glide, and with an active cervical extension.
  Interventions: Procedure: SHAM SNAG
- CONTROL GROUP (No Intervention): The control group did not receive any type of intervention, they only waited for four minutes, sat down on a chair

INTERVENTIONS:
Procedure: sustained natural apophyseal glides — It consists on a sustained apophyseal glides in a postero-anterior direction on C2 with a dose of three series of ten repetitions each
  Other Names: SNAG
  Arms: SNAG GROUP
Procedure: SHAM SNAG — Subjects on SNAG group received a simulation of the contact used for the SNAGs, without any vertebral glide, and with an active cervical extension
  Arms: SHAM SNAG GROUP

SUMMARY:
This analysis aims to evaluate the immediate effect that cervical sustained natural apophyseal glides (SNAGs) have on a group of individuals with induced vertigo by a caloric vestibular stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects,
* Age 18-44 years.

Exclusion Criteria:

* Consume of antipsychotics, antidepressants, antiarrythmics and/or anticonvulsivants
* Hippoacusia
* Auditory diseases
* Peripheral or central vestibulopathies
* Cerviogenic dizziness
* Balance disorders
* Nistagmus
* Oculomotor nerve dysfunctions
* Migraine
* Cervical osteoporosis, lashing or fracture
* Discal cervical hernia
* Cervical neuropathy
* Psychriatic disorders
* Epilepsy
* Pregnancy

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-03 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
vHIT (Video Head Impulse Test) | 15 minutes
  Detection of peripheral vestibular deficits and their recovery

SECONDARY OUTCOMES:
Anxiety | 5 minutes
  state-trait anxiety was measured at the beginning of the study using the Spanish version of the trait-state anxiety inventory (STAI)

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - CSEU La Salle, Madrid
  - Jose V Leon Hernandez, Madrid

IPD SHARING:
Plan to Share IPD: No
Data will only be treated by study researchers